CLINICAL TRIAL: NCT04610762
Title: Using the Cepheid GeneXpert HCV VL Fingerstick Test as a Diagnostic Tool for Chronic Hepatitis C Among Drug Users in Brussels
Brief Title: HCV RNA Fingerstick Assay as Useful Point of Care of Diagnostic Tool for Drug Users in Brussels
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Cepheid (Industry); Réseau Hépatite C Bruxelles (Unknown); Gilead Sciences (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: CE/20-10-01
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Drug user, Point-of-care of molecular diagnostics, hepatitis C RNA, Fingerstick, GeneXpert HCV Viral Load, linkage to care
MeSH Terms: conditions — Hepatitis C, Chronic; Drug Misuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- (Ex) Drug users recognized at-risk population of infection with Hepatitis C virus
  Interventions: Diagnostic Test: GeneXpert HCV VL Fingerstick test

INTERVENTIONS:
Diagnostic Test: GeneXpert HCV VL Fingerstick test — The participants will have a molecular test (GeneXpert HCV VL Fingerstick, Cepheid) that quantifies hepatitis C virus (HCV) RNA levels directly from a fingerstick blood sample.

SUMMARY:
The main objective of this study is to assess the interest (linkage to care) of the Cepheid GeneXpert HCV VL Fingerstick test in Brussels among drug users or former users in contact with the Réseau Hépatite C Bruxelles organization through different partners of this network.

ELIGIBILITY:
Inclusion Criteria:

* (ex) drug users
* a risk of Hepatitis C infection
* French speaking
* Either patient with a positive serology for HCV who have never performed HCV RNA by Polymerase chain reaction (PCR) by a peripheral venous sampling (due to difficult venous access, financial problem, medical insurance problem or other reasons) either patient with a suspicion of reinfection for whom the HCV RNA PCR by peripheral venous sampling is not reimbursed by health insurance

Exclusion Criteria:

* Age <18 years
* Cepheid GeneXpert HCV VL Fingerstick will not use to assess the Sustained Virological Response (SVR) at 12 weeks after the end of an antiviral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All marginalized (ex) drug users with a positive serology (for HCV) without a confirmed diagnosis of chronic hepatitis C, who are in contact with the Réseau Hépatite C Bruxelles organization and other front-line partners in Brussels
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of interest and impact of this new method by the number of participants tested in outreach approaches | 1 year after the start of recruitment

SECONDARY OUTCOMES:
Acceptability by the participants of the use of the Cepheid GeneXpert HCV VL Fingerstick | on day of enrollment
  The participants will answer to a qualitative questionnaire about the Cepheid device and will give their preference between the Cepheid GeneXpert HCV VL test to routine venous tests
Number of participants with a positive HCV RNA test with Cepheid GeneXpert HCV VL Fingerstick who will be taken in charge by hepatologist | one year after enrollment
Number of participants with a positive HCV RNA test with Cepheid GeneXpert HCV VL Fingerstick who will initiate a anti-viral treatment | one year after enrollment
Number of participants with a positive HCV RNA test with Cepheid GeneXpert HCV VL Fingerstick who have a Sustained Virological Response (SVR) at 12 weeks after the end of treatment | one year after enrollment
Time between a positive HCV RNA test with Cepheid GeneXpert HCV VL Fingerstick and the initiation of antiviral treatment | up one year after enrollment
Time between a positive HCV RNA test with Cepheid GeneXpert HCV VL Fingerstick and a recovery defined by a Sustained Virological Response (SVR) | up one year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Mulkay, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre; Lise Meunier, MD, Principal Investigator — ASBL Réseau Hépatite C Bruxelles
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

REFERENCES:
- [Background] Grebely J, Bruneau J, Lazarus JV, Dalgard O, Bruggmann P, Treloar C, Hickman M, Hellard M, Roberts T, Crooks L, Midgard H, Larney S, Degenhardt L, Alho H, Byrne J, Dillon JF, Feld JJ, Foster G, Goldberg D, Lloyd AR, Reimer J, Robaeys G, Torrens M, Wright N, Maremmani I, Norton BL, Litwin AH, Dore GJ; International Network on Hepatitis in Substance Users. Research priorities to achieve universal access to hepatitis C prevention, management and direct-acting antiviral treatment among people who inject drugs. Int J Drug Policy. 2017 Sep;47:51-60. doi: 10.1016/j.drugpo.2017.05.019. Epub 2017 Jul 3. PMID 28683982
- [Background] Day E, Hellard M, Treloar C, Bruneau J, Martin NK, Ovrehus A, Dalgard O, Lloyd A, Dillon J, Hickman M, Byrne J, Litwin A, Maticic M, Bruggmann P, Midgard H, Norton B, Trooskin S, Lazarus JV, Grebely J; International Network on Hepatitis in Substance Users (INHSU). Hepatitis C elimination among people who inject drugs: Challenges and recommendations for action within a health systems framework. Liver Int. 2019 Jan;39(1):20-30. doi: 10.1111/liv.13949. Epub 2018 Sep 22. PMID 30157316
- [Background] Bajis S, Dore GJ, Hajarizadeh B, Cunningham EB, Maher L, Grebely J. Interventions to enhance testing, linkage to care and treatment uptake for hepatitis C virus infection among people who inject drugs: A systematic review. Int J Drug Policy. 2017 Sep;47:34-46. doi: 10.1016/j.drugpo.2017.07.002. Epub 2017 Aug 7. PMID 28797498
- [Background] Chevaliez S, Poiteau L, Rosa I, Soulier A, Roudot-Thoraval F, Laperche S, Hezode C, Pawlotsky JM. Prospective assessment of rapid diagnostic tests for the detection of antibodies to hepatitis C virus, a tool for improving access to care. Clin Microbiol Infect. 2016 May;22(5):459.e1-6. doi: 10.1016/j.cmi.2016.01.009. Epub 2016 Jan 22. PMID 26806260
- [Background] Foucher J, Reiller B, Jullien V, Leal F, di Cesare ES, Merrouche W, Delile JM, de Ledinghen V. FibroScan used in street-based outreach for drug users is useful for hepatitis C virus screening and management: a prospective study. J Viral Hepat. 2009 Feb;16(2):121-31. doi: 10.1111/j.1365-2893.2008.01050.x. Epub 2008 Oct 17. PMID 19175876
- [Background] McHugh MP, Wu AHB, Chevaliez S, Pawlotsky JM, Hallin M, Templeton KE. Multicenter Evaluation of the Cepheid Xpert Hepatitis C Virus Viral Load Assay. J Clin Microbiol. 2017 May;55(5):1550-1556. doi: 10.1128/JCM.02460-16. Epub 2017 Mar 8. PMID 28275079
- [Background] Gupta E, Agarwala P, Kumar G, Maiwall R, Sarin SK. Point -of -care testing (POCT) in molecular diagnostics: Performance evaluation of GeneXpert HCV RNA test in diagnosing and monitoring of HCV infection. J Clin Virol. 2017 Mar;88:46-51. doi: 10.1016/j.jcv.2017.01.006. Epub 2017 Jan 29. PMID 28160728
- [Background] Grebely J, Lamoury FMJ, Hajarizadeh B, Mowat Y, Marshall AD, Bajis S, Marks P, Amin J, Smith J, Edwards M, Gorton C, Ezard N, Persing D, Kleman M, Cunningham P, Catlett B, Dore GJ, Applegate TL; LiveRLife Study Group. Evaluation of the Xpert HCV Viral Load point-of-care assay from venepuncture-collected and finger-stick capillary whole-blood samples: a cohort study. Lancet Gastroenterol Hepatol. 2017 Jul;2(7):514-520. doi: 10.1016/S2468-1253(17)30075-4. Epub 2017 Apr 22. PMID 28442271
- [Background] Yehia BR, Schranz AJ, Umscheid CA, Lo Re V 3rd. The treatment cascade for chronic hepatitis C virus infection in the United States: a systematic review and meta-analysis. PLoS One. 2014 Jul 2;9(7):e101554. doi: 10.1371/journal.pone.0101554. eCollection 2014. PMID 24988388
- [Background] Iversen J, Grebely J, Catlett B, Cunningham P, Dore GJ, Maher L. Estimating the cascade of hepatitis C testing, care and treatment among people who inject drugs in Australia. Int J Drug Policy. 2017 Sep;47:77-85. doi: 10.1016/j.drugpo.2017.05.022. Epub 2017 Jun 1. PMID 28578863
- [Background] Lamoury FMJ, Bajis S, Hajarizadeh B, Marshall AD, Martinello M, Ivanova E, Catlett B, Mowat Y, Marks P, Amin J, Smith J, Ezard N, Cock V, Hayllar J, Persing DH, Kleman M, Cunningham P, Dore GJ, Applegate TL, Grebely J; LiveRLife Study Group. Evaluation of the Xpert HCV Viral Load Finger-Stick Point-of-Care Assay. J Infect Dis. 2018 May 25;217(12):1889-1896. doi: 10.1093/infdis/jiy114. PMID 29534185
- [Background] Bielen R, Koc OM, Busschots D, Verrando R, Nevens F, Robaeys G. Validation of hepatitis C virus RNA detection using capillary blood by finger prick (GenXpert system)-Hepatitis C fingerprick study. J Viral Hepat. 2020 Jul;27(7):709-714. doi: 10.1111/jvh.13284. Epub 2020 Mar 13. PMID 32106345
- [Background] Bajis S, Maher L, Treloar C, Hajarizadeh B, Lamoury FMJ, Mowat Y, Schulz M, Marshall AD, Cunningham EB, Cock V, Ezard N, Gorton C, Hayllar J, Smith J, Whelan M, Martinello M, Applegate TL, Dore GJ, Grebely J; LiveRLife Study Group. Acceptability and preferences of point-of-care finger-stick whole-blood and venepuncture hepatitis C virus testing among people who inject drugs in Australia. Int J Drug Policy. 2018 Nov;61:23-30. doi: 10.1016/j.drugpo.2018.08.011. Epub 2018 Oct 25. PMID 30388566
- [Background] Saludes V, Antuori A, Lazarus JV, Folch C, Gonzalez-Gomez S, Gonzalez N, Ibanez N, Colom J, Matas L, Casabona J, Martro E. Evaluation of the Xpert HCV VL Fingerstick point-of-care assay and dried blood spot HCV-RNA testing as simplified diagnostic strategies among people who inject drugs in Catalonia, Spain. Int J Drug Policy. 2020 Jun;80:102734. doi: 10.1016/j.drugpo.2020.102734. Epub 2020 May 26. PMID 32470849